CLINICAL TRIAL: NCT06675721
Title: A Survey of Acceptance and Factors Associated With Hesitancy Vaccination in a Socioeconomically Disadvantaged Population and Professionals Working in a City Located in Northeast Brazil
Brief Title: A Survey of Acceptance and Factors Associated With Hesitancy Vaccination in Northeast Brazil
Status: Not yet recruiting | Type: Observational
Sponsor: Centro De Estudos E Pesquisas Em Molestias Infecciosas (Other)
Collaborators: MSD Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: EII1001HEVANO
Record Dates: First submitted 2024-08-19; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Vaccine Hesitancy; Vaccine Refusal
MeSH Terms: conditions — Vaccination Hesitancy; Vaccination Refusal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vulnerable group: Individuals who are over 18 years old and are residents of the socioeconomically vulnerable neighborhoods.
  Interventions: Other: Study Questionnaire
- Health Professionals: Healthcare professionals who work in Natal.
  Interventions: Other: Study Questionnaire

INTERVENTIONS:
Other: Study Questionnaire — A survey questionnaire to assess factors related to vaccination adherence, including factors such as vaccine novelty, cost, and prior knowledge among vulnerable populations.

SUMMARY:
The objective of this study is to investigate vaccination acceptance and identify the reasons why people are not vaccinated.

People over 18 years of age who live in neighborhoods with socioeconomic vulnerability and with many cases of infectious diseases, as well as health professionals, will respond to a research questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are over 18 years old and are residents of the PAJUÇARA, FELIPE CAMARÃO, LAGOA AZUL, or PLANALTO neighborhoods, willing to answer the study questionnaire.
* Healthcare professionals who work in Natal, willing to answer the study questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Vulnerable populations residing in neighborhoods characterized by socioeconomic vulnerability and high infectious disease incidence. Four neighborhoods in Natal will be the focus, each with their respective population: Lagoa Azul (61,289), Pajuçara (58,021), Felipe Camarão (50,997), and Planalto (31,206).
  In this project, the inclusion of health professionals as a unified group is essential because of their critical role as trusted source of health information. In Natal, these professionals consist of 5,238 physicians and an estimated 7,066 nurses (derived from a 61.6% prevalence applied to the 11,471 registered nurses in Rio Grande do Norte).
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Resistance to adherence to vaccination | Baseline
  Resistance to adherence to vaccination will be measured using a questionnaire developed for this survey. The questionnaire will be described by mean and standard deviation, and the distribution frequency of each item will be presented, comparing cohorts of health professionals and populations in socioeconomic vulnerability.

CONTACTS AND LOCATIONS:
Overall Officials: Kleber G Luz, PhD, Principal Investigator — Centro De Estudos E Pesquisas Em Molestias Infecciosas

IPD SHARING:
Plan to Share IPD: No